CLINICAL TRIAL: NCT02899780
Title: Treatment of Infected Dialysis Catheters With Fiber Optic Ultraviolet Light
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Ultraviolet Interventions (Industry)
Collaborators: University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UVI-Pilot
Record Dates: First submitted 2016-08-27; First posted 2016-09-14 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Catheter-Related Infections
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Ultraviolet arm (Experimental): This arm will have their dialysis catheters treated with an ultraviolet light emitting optical fiber.
  Interventions: Device: Ultraviolet light emitting optical fiber

INTERVENTIONS:
Device: Ultraviolet light emitting optical fiber — A ultraviolet light emitting optical fiber will be threaded through the existing catheter and withdrawn.
  Other Names: Lumenati Fiber

SUMMARY:
This study is a first-in-man clinical trial using fiber optically delivered ultraviolet light for reducing viable bacteria within indwelling tunneled dialysis catheters.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Have the ability to provide informed consent
* Have an implanted dialysis catheter of one of the following models: Medcomp Titan 15.5F x 24 cm or Medcomp Titan 15.5F x 28 cm
* Positive blood culture drawn from the catheter

Exclusion Criteria:

* Previous inclusion in study
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Quantitative reduction of bacterial counts from blood cultures drawn from the dialysis catheter | Measured immediately after UV treatment
Proportion of patients with any reduction of bacterial counts from blood cultures drawn from the dialysis catheter | Measured at study end, expected at 1 year.

SECONDARY OUTCOMES:
Number of colony forming units (CFU) per cm2 of surface area on the inner lumen of removed catheters | Measured after UV treatment, with results expected in 5 days.
Procedural complications, including excessive bleeding, infection, vascular injury, and significant catheter damage. | Measured at study end, expected at 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Nabeel Akhter, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No